CLINICAL TRIAL: NCT00870779
Title: Co-registered Fluorescence-Enhanced Resection of Brain Tumors Stage I: Correlation With MR and Biopsy
Brief Title: Fluorescence Guided Resection of Brain Tumors
Acronym: FGR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David W. Roberts (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, David W. Roberts, Professor of Surgery (Neurosurgery), Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DMS 0711; R01NS052274-01A2 (NIH)
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Brain Tumors
Keywords: Fluorescence; Brain Tumor; Malignant Glioma; Pituitary Tumor; Skull Base Tumor; Brain Lesions; Brain Metastases; Meningioma
MeSH Terms: conditions — Brain Neoplasms; Glioma; Pituitary Neoplasms; Skull Base Neoplasms; Meningioma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-aminolevulinic acid (Experimental)
  Interventions: Drug: 5-aminolevulinic acid

INTERVENTIONS:
Drug: 5-aminolevulinic acid — 20mg/kg 3 hours prior to surgery
  Other Names: 5-ALA

SUMMARY:
Removing a tumor from your brain is hard to do because, very often, brain tumors do not have boundaries that are easy for your surgeon to find. In many cases, the surgeon can't tell exactly where the tumor begins or ends. The surgeon usually can remove most of your tumor by looking at the MRI images that were taken of your brain before surgery. However, the surgeon does not have any good way to tell if the entire tumor has been removed or not. Removing the entire tumor is very important because leaving tumor behind may allow it to grow back which could decrease your chances of survival.

It is possible to detect tumor cells by making them glow with a specific color of light (a process called fluorescence). This can be done by having you take the drug, ALA, before your surgery. ALA is a molecule that already exists in the cells of your body. Once enough of it is in your body, it gets converted into another molecule named PpIX. If blue light is shined on a tumor that has enough PpIX, it will glow with red light (fluorescence) that can be detected with a special camera. In this study, we want to determine how the fluorescence (red light) is related to the tumor which appears in the images that are normally taken of your brain (which the surgeon uses to guide the removal of your tumor) and the tumor tissue that will be removed during your surgery. Removing the entire tumor is very important because leaving tumor behind may allow it to grow back which could decrease your chances of survival.

DETAILED DESCRIPTION:
The first phase of study (Stage I) will use FI coregistered with pMR, iUS and iSV images to test the overall hypothesis that there is a high degree of spatial correlation between local tissue FI signal and coregistered conventional imaging and corresponding histopathology. Additionally, coregistered probe measurements and biopsy specimens will be acquired intraoperatively. Biopsy specimens will be processed post-operatively (via fluorescence microscopy and chemical spectrofluorimetry) to assess PpIX concentration which will allow direct comparisons of FI signal strength with PpIX production (based on both in vivo probe data and ex vivo histological quantification) as a function of histological grade. The study protocol is outlined below. Because of the overall interest and importance of relating this data to the existing body of literature and the excellent safety record of oral administration of ALA reported in these trials [1, 33-36], we will use the same dose/time schedule described in [1, 33]. The operative procedures will follow existing practice at Dartmouth for image-guided resection of meningiomas, pituitary adenomas and metastases with additional acquisition of FI and biopsy data at predefined time points that are related to the expected volume of tumor tissue. In this first phase of the study, resection decisions will not be made based on FI data alone. Should residual fluorescence remain after the intended resection volume has been removed further excisions will require biopsy confirmation in the OR. It is anticipated that 234 patients will be enrolled in Stage I.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative diagnosis of either presumed low or high grade glioma (astrocytoma, oligodendroglioma, mixed oligo-astrocytoma, anaplastic astrocytoma, and glioblastoma multiforme) or meningioma, pituitary adenoma or metastasis.
* Tumor judged to be suitable for open cranial resection based on preoperative imaging studies.
* Patient able to provide written informed consent.
* Age ≥ 21 years old.

Exclusion Criteria:

* Pregnant women or women who are breast feeding
* History of cutaneous photosensitivity, porphyria, hypersensitivity to porphyrins, photodermatosis, exfoliative dermatitis
* History of liver disease within the last 12 months,
* AST, ALT, ALP or bilirubin levels greater than 2.5 times the normal limit at any time during the previous 2 months
* Plasma creatinine in excess of 180 mol/L.
* Inability to comply with the photosensitivity precautions associated with the study
* Patients with an existing DSM-IV Axis 1diagnosis
* Inability to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-05; Primary Completion 2012-07-02 (Actual); Study Completion 2013-07-02 (Actual)

PRIMARY OUTCOMES:
Determine the degree of spatial correlation between local fluorescence recorded intraop and coregistered conventional imaging obtained preop with MR and intraop with ultrasound and operating microscope stereovision. | From date of first surgery through 6/1/2013

SECONDARY OUTCOMES:
Establish the clinical feasibility of integrating FI with conventional image guidance (pMR, iUS and iSV data). Determine the relationships between FI signals, PpIX concentration, histological grade and image features evident for surgical guidance. | From date of first surgery through 6/1/2013

CONTACTS AND LOCATIONS:
Overall Officials: David W Roberts, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Keith Paulsen, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States